CLINICAL TRIAL: NCT00523406
Title: Comparison of Reduced Fluence Versus Standard Photodynamic Therapy (in Combination With Intravitreal Triamcinolone Acetate)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Stefan Sacu, Assoc. Prof. PD Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EK049/2005
Record Dates: First submitted 2007-08-29; First posted 2007-08-31 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Macular Degeneration
Keywords: choroidal neovascularisation,; vision,; macula,; macular degeneration; optical coherence tomography; neovascular age related macular degeneration
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization | interventions — Photochemotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): standard fluence photodynamic therapy and intravitreal triamcinolone combination
  Interventions: Procedure: Photodynamic therapy and intravitreal triamcinolone
- B (Active Comparator): reduced fluence photodynamic therapy and intravitreal triamcinolone combination
  Interventions: Procedure: Photodynamic therapy and intravitreal triamcinolone

INTERVENTIONS:
Procedure: Photodynamic therapy and intravitreal triamcinolone — combination of photodynamic therapy and intravitreal triamcinolone combination to treat neovascular AMD

SUMMARY:
To assess the CNV treatment effect of PDT with verteporfin in combination with IVTA using reduced fluence compared to the standard fluence.

DETAILED DESCRIPTION:
Age-related macular degeneration (AMD) is by far the most common disorder in the group of irreversible causes of visual disability. AMD leads to dysfunction and loss of photoreceptors in the central retina. Neovascular AMD affects visual function early in the disease process and severely compromises the highly developed functions of the macula, such as perception of details, central fixation, color vision, and reading ability. AMD-related visual impairment is associated with a loss of autonomy and quality of life. Currently, laser photocoagulation, photodynamic therapy (PDT) with verteporfin usually combined with intravitreal triamcinolone acetonide (IVTA) are the only proved treatments for subfoveal choroidal neovascularisation (CNV). Laser photocoagulation is limited to selected cases. Photodynamic therapy using verteporfin provides very promising data regarding improvement of visual acuity and absence of fluorescein leakage. PDT was recently successfully combined with an intravitreal injection of the corticosteroid triamcinolone acetonide. Yet, PDT also leads to damage to surrounding normal choroidal vessels. A pilot trial comparing low fluence (300 mW/cm²) with standard fluence (600 mW/cm²) demonstrated a trend for improved outcomes using the low fluence regimen (VIM study). However, vascular mechanisms and choroidal damage were not examined, and the study group was too small to evaluate vision outcome parameters. Combined with the IVTA, the low fluence effects of PDT may be sufficient for CNV occlusion and the physiological choroids should be spared from any collateral damage. The aim of this study was to compare reduced fluence with standard fluence PDT using verteporfin and IVTA for CNV secondary to AMD.

ELIGIBILITY:
Inclusion criteria:

* Patients 50 years of age or greater.
* Patients with subfoveal choroidal neovascularization lesions secondary to AMD.
* CNV lesion in the study eye is ≤ 4 disc areas in greatest linear dimension.
* Patients who have a BCVA score better than 20/400 in the study eye using ETDRS.
* Only one eye will be assessed in the study. If both eyes are eligible, the one with the worse visual acuity will be selected for treatment and study unless, based on medical reasons, the investigator deems the other eye the more appropriate candidate for treatment and study.

Exclusion Criteria:

* Prior treatment in the study eye with verteporfin, external-beam radiation therapy, subfoveal focal laser photocoagulation, vitrectomy, submacular surgery, or transpupillary thermotherapy.
* Previous or current intravitreal drug delivery (e.g., intravitreal corticosteroid injection or device implantation) in the study eye.
* Laser photocoagulation (juxtafoveal or extrafoveal) in the study eye within one month preceding Visit 1.
* History of glaucoma filtration surgery, corneal transplant surgery or extracapsular extraction of cataract with phacoemulsification within six months preceding Visit 1, or a history of post-operative complications within the last 12 months preceding Visit 1 in the study eye (uveitis, cyclitis etc.).
* History of uncontrolled glaucoma in the study eye (defined as intraocular pressure ≥ 25 mmHg despite treatment with anti-glaucoma mediation).
* Aphakia or absence of the posterior capsule in the study eye.
* Presence of a retinal pigment epithelial tear involving the macula in the study eye.
* Any concurrent intraocular condition in the study eye (e.g., cataract or diabetic retinopathy) that, in the opinion of the investigator, could either require medical or surgical intervention during the three-month study period to prevent or treat visual loss that might result from that condition.
* Active intraocular inflammation (grade trace or above) in the study eye.
* Any active infection involving eyeball adnexa.
* Vitreous hemorrhage or history of rhegmatogenous retinal detachment or macular hole (Stage 3 or 4) in the study eye.
* Ocular conditions that require chronic concomitant therapy with systemic or topical ocular corticosteroids. Chronic concomitant therapy is defined as multiple doses taken daily for three or more consecutive days at any time within six months prior to screening or during the course of the study.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-08; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
• Chorioretinal perfusion. • Perfusion of the neovascular net (CNV). • Changes of intraretinal morphologies. • Central visual function. | one year

SECONDARY OUTCOMES:
macular sensitivity, three dimensional optical coherence tomography | one year

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Schmidt-Erfurth, MD, Prof., Principal Investigator — Department of Ophthalmology, MUVienna
Locations (1):
- Medical University of Vienna, Department of Ophthalmology, Vienna, Austria